CLINICAL TRIAL: NCT01395342
Title: Assessment of Physical Exercise Using Stationary Bicycle for Pregnant Women With Risk for Preeclampsia Development
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Jose Luiz Pinto e Silva, PhD, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08/2011/PC
Record Dates: First submitted 2011-07-04; First posted 2011-07-15 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Pre-eclampsia; Hypertension, Pregnancy-Induced; Pregnancy, High-Risk
Keywords: Pregnant women; Pre-eclampsia; Exercise; Hypertension, Pregnancy-Induced; Parturition
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Motor Activity | interventions — Blood Pressure; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- blood pressure and heart rate data (No Intervention)
  Interventions: Other: Exercise using stationary bicycle

INTERVENTIONS:
Other: Exercise using stationary bicycle — Before exercise, blood pressure and heart rate are measured in the sitting position.
  Exercise is realized using stationary bicycle (horizontal bench mode) once at week, during 20 minutes under physiotherapist supervision.
  The heart rate was maintained at 20% above resting heart rate and up to 140 bpm.
  After exercise is performed a leg stretching and a low back stretching. The blood pressure and heart rate are measured in the sitting position.
  Other Names: incidence of pre-eclampsia; types of birth; perinatal outcomes; blood pressure; heart rate

SUMMARY:
Introduction:

Hypertensive disorders during pregnancy are an important issue in global public health. It is current the leading cause of maternal mortality in Brazil.

Objective:

To assess the effect of physical exercise using stationary bicycle through blood pressure and heart rate measurements, incidence of pre-eclampsia and quality of life survey in pregnant women with chronic high blood pressure, previous preeclampsia pregnancies or both factors associated comparing to a group with no intervention. Verify the type of births, maternal and perinatal outcomes in both groups. Methodology: This randomized clinical trial enrolled pregnant women presenting chronic hih blood pressure, previous pre-eclampsia experience or both. Women from 12 to 20 gestational weeks were selected from the prenatal outpatient clinic and randomly allocated to the study or non-interventional group. Women at the study group performed physical exercise using stationary bicycle (horizontal bench model) during 20 minutes, once a week. The heart rate was maintained at 20% above resting heart rate and up to 140 bpm. Blood pressure and heart rate measurements were evaluated before and after exercise. The non-intervention group followed regular prenatal routine with weekly returns for heart rate and blood pressure measurements. Both groups fulfilled the quality of life survey (SF-36 questionnaire) at three times: between 12 and 20 weeks; 28 and 32 weeks and 36 and 41 weeks of gestation. After that data of parturition will be analyzed to compare the incidence of pre-eclampsia, types of birth, maternal and perinatal outcomes.

DETAILED DESCRIPTION:
Significance was assumed as p<.5%.

ELIGIBILITY:
Inclusion Criteria:

* pregnant with 12 to 20 weeks gestational
* have chronic blood pressure, previous pre-eclampsia or both
* able to perform a exercise

Exclusion Criteria:

* multiple pregnancy
* Systemic lupus erythematosus
* heart disease
* neurological disease
* renal failure
* persistent vaginal bleeding
* isthmic-cervical insufficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Risk to development pre-eclampsia | up to 28 weeks
  The comparison between groups will be by the diagnosis of pre-eclampsia. Pre-eclampsia is diagnosed after 20 week of gestation with systolic blood pressure equal to or greater than 140 mmHg, diastolic blood pressure equal to or greater than 90 mmHg and proteinuria greater than or equal 0.3 g/d by 24 hour urine collection.

SECONDARY OUTCOMES:
Types of birth | up to 28 weeks
  Parturition data will be analyzed.
Perinatal outcomes | up to 28 weeks
  Number of participants with adverse events. Prematurity by CAPURRO method, APGAR score to measure the health of newborn.

CONTACTS AND LOCATIONS:
Overall Officials: João Luiz C Pinto e Silva, Study Director — University of Campinas (Unicamp)
Locations (1):
- Hospital da Mulher Professor Doutor José Aristodemo Pinotti - CAISM/UNICAMP, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Kasawara KT, Burgos CS, do Nascimento SL, Ferreira NO, Surita FG, Pinto E Silva JL. Maternal and Perinatal Outcomes of Exercise in Pregnant Women with Chronic Hypertension and/or Previous Preeclampsia: A Randomized Controlled Trial. ISRN Obstet Gynecol. 2013 Aug 12;2013:857047. doi: 10.1155/2013/857047. eCollection 2013. PMID 23997960